CLINICAL TRIAL: NCT06522828
Title: A Phase 2 Study to Evaluate the Safety and Efficacy of SSGJ-707 in Advanced Gynecologic Cancer Patients
Brief Title: A Study to Evaluate SSGJ-707 in Advanced Gynecologic Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSGJ-707-ST-II-02
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Advanced/recurrent Endometrial Cancer and Platinum-resistant Ovarian Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- SSGJ-707(dose 1)+ carboplatin + paclitaxel (Experimental)
  Interventions: Drug: SSGJ-707; Drug: carboplatin; Drug: paclitaxel
- SSGJ-707(dose 2)+ carboplatin + paclitaxel (Experimental)
  Interventions: Drug: SSGJ-707; Drug: carboplatin; Drug: paclitaxel
- SSGJ-707(dose 3)+ carboplatin + paclitaxel (Experimental)
  Interventions: Drug: SSGJ-707; Drug: carboplatin; Drug: paclitaxel
- SSGJ-707(dose 4)+ paclitaxel (Experimental)
  Interventions: Drug: SSGJ-707; Drug: paclitaxel

INTERVENTIONS:
Drug: SSGJ-707 — SSGJ-707 is a bispecific antibody against human PD-1 and VEGF
Drug: carboplatin — chemotherapy
  Arms: SSGJ-707(dose 1)+ carboplatin + paclitaxel; SSGJ-707(dose 2)+ carboplatin + paclitaxel; SSGJ-707(dose 3)+ carboplatin + paclitaxel
Drug: paclitaxel — chemotherapy

SUMMARY:
This is an open, multicenter Phase II clinical study of SSGJ-707 combined with chemotherapy in the treatment of advanced/recurrent endometrial cancer and platinum-resistant ovarian cancer. The objective is to evaluate the safety, tolerability and antitumor activity of SSGJ-707 in the treatment of advanced/recurrent endometrial cancer and platinum-resistant ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-75 years old
2. Advanced endometrial cancer and platinum-resistant ovarian cancer
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Expected survival >=12 weeks.
5. Signed informed consent form.

Exclusion Criteria:

1. Known uncontrolled or symptomatic central nervous system metastatic disease.
2. Adverse events (with exception of alopecia and fatigue) from any prior anticancer therapy of grade >1 (National Cancer Institute Common terminology Criteria [NCI CTCAE] v.5.0).
3. Inadequate organ or bone marrow function.
4. Pregnant or breast-feeding woman.
5. Known allergies, hypersensitivity, or intolerance to SSGJ-707 The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
ORR | 12 months
  Objective response rate
Safety and tolerability | 12 months
  Safety and tolerability assessed by incidence and severity of adverse events

SECONDARY OUTCOMES:
PFS | 24 months
  The efficacy end point

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing Cancer Hospital, Chongqing, China

IPD SHARING:
Plan to Share IPD: No